CLINICAL TRIAL: NCT00023959
Title: A Phase I Study Of Bevacizumab (Recombinant Humanized Monoclonal Antibody To Vascular Endothelial Growth Factor) In Addition To Flourouracil And Hydroxyurea As Initial Chemotherapy With Concomitant Radiotherapy (B-FHX) For Poor Prognosis Head And Neck Cancer
Brief Title: Bevacizumab, Fluorouracil, and Hydroxyurea Plus Radiation Therapy in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02408; 11033B; CDR0000068879 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Basal Cell Carcinoma of the Lip; Stage III Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage III Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Lymphoepithelioma of the Oropharynx; Stage III Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Hydroxyurea; Fluorouracil; Bevacizumab; Radiotherapy; Radiation; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (hydroxyurea, fluorouracil, bevacizumab, radiation) (Experimental): Patients receive oral hydroxyurea every 12 hours on days 1-6, fluorouracil IV continuously on days 1-5, and bevacizumab IV over 90 minutes on day 1. Patients also undergo radiotherapy once daily on days 1-5. Patients receive G-CSF subcutaneously on days 6-12. Treatment repeats every 2 weeks for up to 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: hydroxyurea; Drug: fluorouracil; Biological: bevacizumab; Radiation: radiation therapy; Biological: filgrastim; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: hydroxyurea — Given orally
  Other Names: HU; HYD; Hydrea; Hydroxycarbamide; Hydurea
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining monoclonal antibody therapy with chemotherapy and radiation therapy may be an effective treatment for head and neck cancer. This phase I trial is to see if combining bevacizumab, fluorouracil, and hydroxyurea with radiation therapy works in treating patients who have advanced head and neck cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicity of bevacizumab when given in combination with fluorouracil, hydroxyurea, and radiotherapy in patients with advanced head and neck cancer.

II. Determine the time to progression, pattern of failure, local control, and distant failure rate in patients treated with this regimen.

III. Determine the local toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of bevacizumab.

Patients receive oral hydroxyurea every 12 hours on days 1-6, fluorouracil IV continuously on days 1-5, and bevacizumab IV over 90 minutes on day 1. Patients also undergo radiotherapy once daily on days 1-5. Patients receive filgrastim (G-CSF) subcutaneously on days 6-12. Treatment repeats every 2 weeks for up to 7 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 27-39 patients will be accrued for this study within 5.4-19.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced head and neck cancer

  * Requiring regional palliative radiotherapy
  * Not amenable to standard therapy
* Previously untreated disease allowed only if prognosis is poor (i.e., estimated 2-year survival of less than 10% if treated with standard therapy alone)
* No obvious tumor involvement of major vessels on CT scan
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of bleeding diathesis
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Urine protein no greater than trace
* Urine protein less than 0.5 g/24 hours
* No significant renal impairment
* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No deep venous thrombosis
* No uncontrolled hypertension
* No clinically significant peripheral artery disease
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* No hemoptysis of at least 1 tablespoon
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or other agents used in this study
* No non-healing wounds within the past 4 weeks
* No significant ongoing or active infection
* No other uncontrolled illness
* No other severe complicating medical illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior fluorouracil and hydroxyurea with radiotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* See Disease Characteristics
* See Chemotherapy
* At least 4 months since prior radiotherapy and recovered
* At least 4 weeks since prior major surgery
* No prior or concurrent chronic use of aspirin or other nonsteroidal anti-inflammatory agents
* No other concurrent investigational agents
* No concurrent anticoagulation therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2001-07; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity assessed using NCI CTCAE version 3.0 | 14 weeks

SECONDARY OUTCOMES:
Objective response rate (CR+PR) assessed using RECIST criteria | Up to 9 years
  The associated 95% confidence interval will be determined.
Pattern of failure, described as locoregional, distant, or both | Up to 9 years
Duration of response | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 9 years
Progression free survival | From the date of registration to the date of progressive disease or death, assessed up to 9 years
  Will be calculated using the Kaplan-Meier method, and median progression-free and overall survival times, along with their 95% confidence intervals, will be derived using the procedure described in Brookmeyer and Crowley.
Overall survival | From the date of registration to the date of death, assessed up to 9 years
  Will be calculated using the Kaplan-Meier method, and median progression-free and overall survival times, along with their 95% confidence intervals, will be derived using the procedure described in Brookmeyer and Crowley.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States